CLINICAL TRIAL: NCT05527548
Title: The Effect of Oral Administration of Alendronate on Knee Functions Following Anterior Cruciate Ligament Reconstruction - A Pilot Study of Single-Blind Randomized Controlled Trial
Brief Title: A Single-blind RCT to Investigate the Effect of Alendronate on Knee Function Following ACLR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Pauline Lui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.346
Record Dates: First submitted 2022-09-01; First posted 2022-09-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: ACL Reconstruction
MeSH Terms: interventions — Alendronate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALN group (Experimental): Patients receive weekly dose of 70mg of ALN and a standard rehabilitation program
  Interventions: Drug: Alendronate (ALN)
- Untreated group (No Intervention): Patients receive a standard rehabilitation program

INTERVENTIONS:
Drug: Alendronate (ALN) — The oral ALN is the first-line therapy for osteoporosis, and it has been proven that once-weekly ALN 70 mg is an effective and well-tolerated dose for the treatment of postmenopausal osteoporosis. In this study, after receiving the approval of CREC and the Department of Health, we will purchase ALN from drug store. Previous clinical studies have shown that oral administration of ALN at 70mg/week for 1 year and at 5mg/day for 2 years reduced bone loss in postmenopausal women and patients who underwent total hip arthroplasty, respectively. Therefore, in the proposed study, ALN at the dose of 70mg/week will be given to patients post-ACLR for a duration of 8 weeks.
  Arms: ALN group

SUMMARY:
Anterior cruciate ligament (ACL) is the key ligament connecting the femur to tibia that helps stabilising the knee joint. ACL tear is common. It accounts for over 50% of all knee injuries and affects more than 200,000 people in the United States each year. Patients with ACL tear have a higher risk of developing post-traumatic osteoarthritis. ACL reconstruction (ACLR) with the attachment of tendon grafts within bone tunnels are commonly performed to restore the stability of the joint and thereby minimise injury to both the chondral surface and surrounding tissues. About 130,000 ACLR was performed in the United States in 2006. Both the incidence rates of ACL injuries and ACLR are on the rise, particularly in children and adolescents. Conventional ACLR is not a universally successful procedure, with long healing time and high rates of graft failure (2.8%) and graft laxity (18%). The average cost of an ACLR in the United States was about USD 24,707 ±15,644. The cost for revision surgery and societal cost due to absence from work and sport are expected to be even higher. The demand for a better intervention to improve the outcomes after ACLR and reduce the healing time is huge.

ALN was chosen for the pilot study because it is the most studied BPs, with high bone-binding affinity and more prolonged duration of action. As a member of amino BPs, it also has higher anti-resorptive activities compared to non-amino BPs. Our encouraging results on ALN in the animal studies also provide evidence to support the trial of ALN in human.

ALN have been shown to have a very good safety and tolerability profile. The common side effects of ALN are stomach pain, constipation, diarrhoea, gas, or nausea. Oral ALN seems can induce mild gastro-intestinal disturbances. However, two studies, with subjects treated with ALN for 10 months and 2.9 years, respectively, showed that ALN was not associated with any increased incidence of upper GI tract events. The serious adverse event, oesophageal cancer, has been associated with ALN. However, two published papers with long term observations of 9 and 4.5 years, respectively, showed that ALN was not significantly associated with incident oesophageal or gastric cancer compared with the control group.

This study aims to evaluate the effects of oral administration of ALN on knee stability (primary), peri-tunnel bone loss, tunnel bone formation, knee laxity, knee muscle strength as well as self-reported knee symptoms, function and sports activity over 12 months in patients undergoing ACLR in a pilot study of single-blind randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female with age 18-40 at the time of surgery
* First ACLR
* Single leg involvement
* Able to attend pre-operative assessment
* Voluntarily agreed to participate and signed the informed consent form

Exclusion Criteria:

* Known chronic disease or receiving long-term medications affecting bone metabolism including BPs
* Contraindication to alendronate therapy such as poor dental fitness
* ACL injury less than 6 weeks
* Injury on duty cases
* Patients who have undergone arthroscopy or open surgery in the index knee in the last 12 months
* Other associated injuries (fractures and other ligament involvement such as neurovascular bundles injury)
* Chondral lesion with concomitant intervention
* Presence of X-ray features of osteoarthritis including decrease in joint space, presence of osteophytes and subchondral cysts
* Neurological deficit
* Pregnant or breastfeeding
* Inability to give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Single-leg Hop Test (SLH) | Change from baseline SLH at 8 weeks
  SLH test measures the functional stability of the knee with high intraclass correlation coefficients ranging from 0.97 to 0.99 (59). The patient will be asked to perform single-leg hop on both the injured and non-injured legs three times and the hop distance will be recorded. An index score, calculated by dividing the averaged hop distances of the injured leg by that of the non-injured leg, will be reported.
Single-leg Hop Test (SLH) | Change from baseline SLH at 2 months
  SLH test measures the functional stability of the knee with high intraclass correlation coefficients ranging from 0.97 to 0.99 (59). The patient will be asked to perform single-leg hop on both the injured and non-injured legs three times and the hop distance will be recorded. An index score, calculated by dividing the averaged hop distances of the injured leg by that of the non-injured leg, will be reported.
Single-leg Hop Test (SLH) | Change from baseline SLH at 4 months
  SLH test measures the functional stability of the knee with high intraclass correlation coefficients ranging from 0.97 to 0.99 (59). The patient will be asked to perform single-leg hop on both the injured and non-injured legs three times and the hop distance will be recorded. An index score, calculated by dividing the averaged hop distances of the injured leg by that of the non-injured leg, will be reported.
Single-leg Hop Test (SLH) | Change from baseline SLH at 10 months
  SLH test measures the functional stability of the knee with high intraclass correlation coefficients ranging from 0.97 to 0.99 (59). The patient will be asked to perform single-leg hop on both the injured and non-injured legs three times and the hop distance will be recorded. An index score, calculated by dividing the averaged hop distances of the injured leg by that of the non-injured leg, will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong